CLINICAL TRIAL: NCT05266950
Title: First-in-Human (FIH), Open-Label, Non-Randomized, Single-Arm Phase 1 Study to Evaluate the Safety and Efficacy of CI-135 CAR-T Cells in Subjects with Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Safety and Efficacy Study of CI-135 CAR-T Cells in Subjects with Relapsed or Refractory Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty in joining the group
Sponsor: Beijing Boren Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRYY-IIT-LCYJ-2021-018
Record Dates: First submitted 2021-12-29; First posted 2022-03-04 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: CAR-T; Leukemia; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CI-135 CAR-T (Experimental): chimeric antigen receptor T cell treatment
  Interventions: Biological: CI-135 CAR-T cells (0.5 x 10^6 CAR-T+ cells/kg，1.0 x 10^6 CAR-T+ cells/kg)

INTERVENTIONS:
Biological: CI-135 CAR-T cells (0.5 x 10^6 CAR-T+ cells/kg，1.0 x 10^6 CAR-T+ cells/kg) — Recommended lymphodepletion regimen: cyclophosphamide (250 mg/m2/d, ×3d) and fludarabine (30 mg/m2/d, ×3d). If the patient has a hematological toxicity of grade 3 or higher, the alternative regimen is: cyclophosphamide (125mg/m2/d, ×3d) and fludarabine (15 mg/m2/d, ×3d). During lymphodepletion, physicians can give anti-myeloid drugs such as demethoxydaunorubicin or daunorubicin as appropriate.

SUMMARY:
This is a FIH, single center, open label, non-randomized, single-arm, Phase I clinical trial to evaluate the safety and efficacy of CI-135 CAR-T cells in subjects with relapsed or refractory Acute Lymphoblastic Leukemia. This study is a dose-escalation study that includes 2 dose levels, and a total of 4-7 subjects will be enrolled. CI-135 CAR-T cells will be manufactured using PBMC collected from the subjects, and will be infused intravenously into subjects after lymphodepletion.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥5 years old and ≤70 years old, male or female;
2. Expected survival exceeds 12 weeks;
3. Diagnosed as primary or secondary AML patients that meet the World Health Organization (WHO) classification, and meet any of the following conditions: a) AML patients who have not reached complete remission after at least 3 cycles of standard induction chemotherapy B) AML patients who have achieved complete remission after induction chemotherapy and relapse within 1 year; c) AML patients who have relapsed after achieving complete remission after induction chemotherapy for more than 1 year and have not remitted after 1 course of induction chemotherapy; d) AML patients who have relapsed after transplantation ; E) AML patients who have experienced 2 or more relapses. For patients who meet one of a), b), and c) and have FLT-3 mutations, in addition to induction therapy, they should also receive at least one TKI treatment and has not achieved complete remission or relapsed after complete remission (except patients who cannot tolerate TKI treatment or have contraindications to TKI treatment).
4. The FLT-3 mutation is positive by the leukemia cell gene detection, or the FLT-3 expression is ≥35%;
5. ECOG score 1-2;
6. Liver, kidney, heart and lung functions meet the following requirements:

   1. Glomerular filtration rate ≥60 ml/min/1.73 m2 or serum creatinine ≤2 times the upper limit of normal;
   2. Serum AST, ALT≤3 times the upper limit of normal, and total bilirubin≤1.5 times the upper limit of normal;
   3. Blood oxygen saturation> 92%;
   4. The ventricular ejection fraction ≥50%, there is no pericardial effusion detected by ultrasound, and no clinically significant ECG changes.
7. Able to understand this experiment and sign the informed consent form.

Exclusion Criteria:

1. Diagnosed as acute promyelocytic leukemia (APL M3);
2. Accompanied with other uncontrolled malignant tumors (except those that would not interfere with the safety or efficacy evaluation of the trial).
3. Have received CAR-T cell or other genetically modified cell therapy in the past;
4. Medical history or evidence of significant cardiovascular risk, including any of the following conditions: congestive heart failure, unstable angina, clinically significant arrhythmia (such as ventricular fibrillation, ventricular tachycardia, etc.), performed coronary angioplasty 6 months before infusion, intracardiac defibrillator or any clinically-related complications that may pose a risk to the safety of the subject or interfere with the evaluation, procedures or completion of the research;
5. Subjects who are positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and whose peripheral blood HBV DNA titer test is greater than or equal to the lower limit of detection; those who are positive for hepatitis C virus (HCV) antibody and positive for peripheral blood HCV RNA; Human immunodeficiency virus (HIV) antibody positive; syphilis test positive;
6. Acute or chronic hepatitis C is positive. Exceptions: acute hepatitis C with complete clearance of the virus; chronic hepatitis C, with a sustained virological response 24 weeks after completion of hepatitis C treatment (SVR24) determined an undetectable viral load;
7. A history of arterial or venous thrombosis within 3 months before enrollment;
8. Any graft-versus-host disease that requires systemic application of immunomodulators;
9. A history of central nervous system disease or subjects who need treatment (for example, uncontrolled seizures);
10. Active infection that cannot be controlled.
11. Subjects who are known to be allergic to the components of CI-135 CAR-T cells or any components of the lymphodepletion regimen (cyclophosphamide and fludarabine).
12. Women who are pregnant or breastfeeding, and female patients who plan to become pregnant within 1 year after cell infusion, or male patients whose partners plan to become pregnant within 1 year after their infusion.
13. Other situations that are considered to be unsuitable to participate in the study by researchers.

Ages: 5 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 28 days post intravenous infusion
  Dose-limiting toxicity (DLT)

SECONDARY OUTCOMES:
Adverse events | until two years after cell infusion
  Incidence and severity of adverse events as assessed by NCI-CTCAE 5.0
Concentration of PK CAR positive T cells in peripheral blood | until two years after cell infusion
  PK CAR positive T cells in peripheral blood, PK CAR transgene levels in peripheral blood
Pharmacodynamic data in peripheral blood | until two years after cell infusion
  Time profile of CAR positive T cells concentrations in peripheral blood
Objective response rate (ORR) | until two years after cell infusion
  Objective response rate (ORR)
Duration of remission (DOR) after infusion | until two years after cell infusion
  refers to the time from the first assessment of CR or PR to the first assessment of disease progression or death from any cause
Progression-free survival (PFS) after infusion | until two years after cell infusion
  refers to the time from cell infusion to the first assessment of tumor progression or recurrence or death from any cause
Overall survival (OS) after infusion | until two years after cell infusion
  efers to the time from cell infusion to death due to any cause. For subjects who have dropped out before death, the dates of their last visit would be counted as their time of death; if the subject receives other new treatments, the time of death will be calculated based on the start date of the new treatment; if the study ends, the time of death will be calculated based on the end date
Time of human anti-mouse antibody production persist in human body （Immunogenicity） | until two years after cell infusion
  Immunogenicity will be analyzed during the study, including the time of human anti-mouse antibody production and how long will it last in the body.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Pan, MD/PhD, Principal Investigator — Beijing Gaobo Boren Hospital
Locations (1):
- Beijing Gaobo Boren Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No